CLINICAL TRIAL: NCT05425901
Title: Preclinical Evaluation of Multimodal Therapeutic Strategies in Intestinal Irradiation and Inflammatory Bowel Disease From Organoids
Acronym: INTRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C20-53; 2021-A02973-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Radiation Enteritis; Inflammatory Bowel Diseases
Keywords: colonoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBD (Experimental): active or quiescent
  Interventions: Other: biopsy
- control (Active Comparator): polyp screening
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — endoscopy biopsies (6)

SUMMARY:
This study is carried out in patients with IBD and healthy subjects requiring ileocolonoscopy as part of routine care (disease monitoring or polyp/colon cancer screening). It aims the generation and culturing of organoids from digestive biopsies recovered from healthy and/or pathological (inflammatory) ileal and/or colonic mucosa during an ileo-colonoscopy. These cultures will make it possible to validate the organoid production method used in the context of the research (primary objective). In a second phase (secondary objectives), the study will aim to setup a screening tool by irradiating the organoids (step one) and then evaluate in vitro the regenerative activity of treatments dedicated to improve inflammatory bowel diseases and acute radiation enteritis (step two).

ELIGIBILITY:
Inclusion criteria:

- Group 1: active IBD

* 18 years old or older
* Assured IBD diagnosis (Crohn's disease/ulcerative colitis) according to European Crohn's and Colitis Organisation (ECCO) 2019 consensus criteria
* Active IBD (Harvey-Bradshaw score of 4 or above for Crohn's disease or partial Mayo score of 3 or above for ulcerative colitis)
* Indication to perform a coloscopy
* Written consent for study participation obtained

Or

- Group 2: inactive IBD

* 18 years old or older
* Assured IBD diagnosis (Crohn's disease/ulcerative colitis) according to ECCO 2019 consensus criteria
* Inactive IBD (Harvey-Bradshaw score below 4 for Crohn's disease or partial Mayo score below 3 for ulcerative colitis)
* Indication to perform a coloscopy
* Written consent for study participation obtained

Or

- Group 3: Control

* 18 years old or older
* Indication to perform a coloscopy to detect polyp
* No known bowel disease
* Written consent for study participation obtained

Exclusion Criteria:

* Inability to understand, read, sign informed consent and/or express consent
* Person subject to legal protection (curator, guardianship or safeguard of justice),
* Deprivation of liberty by judicial or administrative decision,
* Non-affiliation to a social security scheme or non-beneficiary of such a scheme
* Pregnant, parturient, breastfeeding women
* Contraindication to performing biopsies
* Participation in other therapeutic research that may modify the behavior of intestinal cells (for example, drug research for the treatment of IBD)
* Anticoagulant treatment or bleeding disorder
* Person subject to a judicial safeguard measure
* People hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Validation of organoid-production method - quantity | Day 1
  Quantity of organoids created
Validation of organoid-production method - size | Day 1
  Size of organoids created
Validation of organoid-production method - cell growth | Day 1
  Cell-growth kinetics
Validation of organoid-production method - cell composition | Day 1
  Cell composition assessed by immunofluorescence
Validation of organoid-production method - cell composition | Day 1
  Cell composition compared to native-biopsy cell composition assessed by single-cell RNA sequencing
Validation of organoid-production method - cell apoptosis | Day 1
  Cell-apoptosis level assessed by immunofluorescence
Validation of organoid-production method - tight junctions | Day 1
  Number of tight junctions between cells assessed by immunofluorescence

SECONDARY OUTCOMES:
Screening-tool setup - quantity | Day 1
  Quantity of organoids after irradiation
Screening-tool setup - size | Day 1
  Size of organoids after irradiation
Screening-tool setup - cell growth | Day 1
  Cell-growth kinetics after irradiation
Screening-tool setup - cell composition | Day 1
  Cell composition after irradiation assessed by immunofluorescence
Screening-tool setup - cell apoptosis | Day 1
  Cell-apoptosis level after irradiation assessed by immunofluorescence
Screening-tool setup - tight junctions | Day 1
  Number of tight junctions between cells after irradiation assessed by immunofluorescence
Screening-tool setup - inflammatory cytokines | Day 1
  Level of inflammatory-cytokines produced after irradiation assessed by single-cell RNA sequencing
In-vitro treatment evaluation - quantity | Day 1
  Quantity of organoids after irradiation and in presence of treatment
In-vitro treatment evaluation - size | Day 1
  Size of organoids after irradiation and in presence of treatment
In-vitro treatment evaluation - cell growth | Day 1
  Cell-growth kinetics after irradiation and in presence of treatment
In-vitro treatment evaluation - cell composition | Day 1
  Cell composition after irradiation and in presence of treatment assessed by immunofluorescence
In-vitro treatment evaluation - cell composition | Day 1
  Cell composition compared to native-biopsy cell composition assessed by single-cell RNA sequencing
In-vitro treatment evaluation - cell apoptosis | Day 1
  Cell-apoptosis level after irradiation and in presence of treatment assessed by immunofluorescence
In-vitro treatment evaluation - tight junction | Day 1
  Number of tight junctions between cells after irradiation and in presence of treatment assessed by immunofluorescence
In-vitro treatment evaluation - inflammatory cytokines | Day 1
  Level of inflammatory-cytokines produced after irradiation and in presence of treatment assessed by single-cell RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Ambroise Paré Hartmann, Neuilly-sur-Seine, Hauts-de-Seine, France